CLINICAL TRIAL: NCT06206694
Title: Serum YKL-40 Levels is Associated With Nutritional and Oxidative Status of Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 112049
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Malnutrition; Oxidative Stress
Keywords: YKL-40; nutrition status; hemodialysis patients; inflammation
MeSH Terms: conditions — Malnutrition; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background

YKL-40 is a glycoprotein that had been reported to be associated with inflammation atherosclerosis and endothelial dysfunction. The objective is to explore the association of serum YKL-40 levels with nutrition status, inflammation, and body composition in a cohort of hemodialysis patients

Methods

We plan to recruit 400 prevalent HD patients. Their baseline serum YKL-40 levels, body anthropometry, the profile of insulin resistance, bioimpedance spectroscopy parameters, and nutritional indices will be measured.

DETAILED DESCRIPTION:
Study Design and Patients

Patients This is a prospective observational study. The patients will be recruited from HD patients at dialysis units of Tungs Taichung Metroharbour Hospital, which is an outpatient facility. The study inclusion criteria of participants are those maintain on HD therapy for at least 3 months prior to enrollment and being in stable condition without co-morbidities such as heart failure, infection, cirrhosis, respiratory disease, nephrotic syndrome, malignancy, chronic liver disease, or severe inflammation. None of the patients are receiving surgical operations or hospitalized in recent 3 months. In this study, written informed consent will be obtained from all participants. The study protocol will be send to the institutional review board of Tungs Taichung Metroharbour Hospital for approval. The study will be registered to the ClinicalTrial. Gov. Registry and will fully adhered to the guidelines of the Declaration of Helsinki

Methodology

Laboratory measurements Blood samples will be collected before dialysis session. Serum biochemistry such as albumin, urea nitrogen, uric acid, creatinine, total cholesterol, triacylglycerol levels, total ion binding capacity (TIBC), 25-hydroxyvitamin D, hemoglobin, and white blood count are measured employing standard laboratory techniques with the use of an automatic analyzer. Serum prealbumin and high-sensitivity C-reactive protein (hs-CRP) are quantified by nephelometry. YKL-40 and interleukin-6 (IL-6) were quantified by a double-sided sandwich-type enzyme-linked immunosorbent assay (ELISA) kit (R&D Systems ; Minneapolis, MN, USA).

Fasting glucose levels were measured, after overnight fast and classified according to the American Diabetes Association (ADA) standards [29]. In addition, the serum insulin level, and hemoglobin A1c level are measured. The assessment of insulin resistance is done using the HOMA-IR index [30]: HOMA - IR = fasting glucose (in mmol/l) × fasting insulin (in µU/ml) / 22.5 Serum insulin, vaspin, and adiponectin level is measured by a commercially available ELISA kit following the manufacturer's instructions. Markers of oxidative stress such as total antioxidant capacity [TAC]), serum advanced oxidation protein products (AOPP) and serum CML (a component of AGEs) will also be measured.

Evaluation of nutritional status and body composition

Anthropometric measures including body weight, body mass index (BMI), waist and hip circumference, mid-arm circumference, and the waist-hip ratio (WHR) will be obtained. BMI is determined by the standard formula and further categorized according to the Asia Pacific version of the WHO classification [31-32]. According to this system, BMI<18 kg/m2 is underweight; 18 to 22.9 is normal weight; 23 to 24.9 is marginal overweight; 25 to 29.9 is overweight; and greater than 30 is obesity [27, 28]. Lastly, the conicity index at baseline is determined to quantify the degree of central obesity [33].

Patients' nutrition status is determined by their serum albumin and pre-albumin levels, Subjective Global Assessment (SGA) score, normalized protein nitrogen appearance (NPNA), and fat-free edema-free body mass (FEBM). The 4-item 7-point SGA scoring system is employed [34]. NPNA was calculated using the modifed Bergstrom's formula [35]. FEBM was calculated using the creatinine kinetic method following the Forbes and Brunining formula [36], and reported as a percentage of their ideal body weight.

We use the multi-frequency bio-impedance spectroscopy device (Body Composition Monitor, Fresenius Medical Care, Germany) as described previously [36, 37]. In this study, the data on lean tissue mass (LTM), adipose tissue mass (ATM), the volume of over-hydration (OH), and the extracellular-tointracellular volume (E: I) ratio will be analyzed.

Statistical analysis All variables were analysed using a Kolmogorov-Smirnov test to classify them as normally or non-normally distributed. Values are given as mean [standard deviation (SD)] or median (IQR). Univariate analysis is performed to examine the relationships between YKL-40 and other parameters employing Spearman's rank correlation coefficient. Multivariate analysis is performed for parameters showing significant differences. Potential confounding factors for increased YKL-40 are assessed using a multiple regression analysis model based on general variables, inflammatory markers and correlations with malnutrition (p<0.10). Two-sided P values of <0.05 are considered to be statistically significant in all analyses. All statistical analyses were performed with the SPSS 23.0 statistical package (SPSS, Chicago, IL, USA). A p-value <0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes aged 20 years or over
* Received stable hemodialysis at least 3 months.
* Written informed consent.

Exclusion Criteria:

* heart failure
* infection
* cirrhosis
* respiratory disease
* nephrotic syndrome
* malignancy
* chronic liver disease
* severe inflammation
* None of the patients are receiving surgical operations or hospitalized in recent 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients have to be at least 20-years-old and hemodialysis (HD) for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Analysis of biomarkers of YKL40 | 1 years
  YKL40 is also reportedly useful as an inflammation marker in HD patients
Evaluation of nutritional status and body composition | 1 years
  Malnutrition, with a prevalence between 40% and 75% in maintenance hemodialysis patients is the most important risk factor for morbidity, the quality of life, all-cause mortality and cardiovascular mortality.

SECONDARY OUTCOMES:
Analysis of biomarkers of IL-6 | 1 years
  The IL-6 was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
vaspin | 1 years
  The vaspin was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
insulin | 1 years
  The insulin was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
adiponectin | 1 years
  The adiponectin was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
total antioxidant capacity | 1 years
  Total antioxidant capacityassay is useful to assay antioxidant levels in serum
AOPP | 1 years
  The IL-6 was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods
Nε-Carboxymethyllysine (CML) | 1 years
  The Nε-Carboxymethyllysine (CML) was determined from plasma samples using standardized enzymelinked immunosorbent assay (ELISA) methods

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided